CLINICAL TRIAL: NCT06675786
Title: The Effect of Catheter Protector on Catheter Dwell Time and Complications in Patients with Peripheral Venous Catheter in the Oncology Clinic
Brief Title: The Effect of Catheter Protector on Catheter Dwell Time and Complications
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karamanoğlu Mehmetbey University (Other)
Responsible Party: Principal Investigator, Tuğba DOST, Principal Investigator, Karamanoğlu Mehmetbey University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Karamanoğlu Mehmetbey üni
Record Dates: First submitted 2024-10-14; First posted 2024-11-05 (Actual); Last update posted 2024-11-05 (Actual); Status verified 2024-10

CONDITIONS: Peripheral Catheterization; Complications
Keywords: Peripheral Venous Catheterization; IV House; Complication; Phlebitis
MeSH Terms: conditions — Phlebitis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Patients will be informed about the study and their consent will be obtained without revealing which group they are in.
  A blind technique will also be applied in terms of statistical analysis in the study. Data will be recorded on the computer as Group A and Group B by the researcher without using the terms experimental and control group. Data analyses will be performed by a statistician other than the person who performed the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- I.V. House UltraDressing (Experimental): The nurse who will perform the PVC will clean the area where the PVC will be applied with alcohol and cotton wool, let it dry and apply Teflon Introcan Safety I.V. Catheter No. 22-24 (B. Braun Medical Inc. Bethlehem, PA, USA) to the patients and apply the routine intravenous line fixation method of the clinic with a plaster. The patient with the PVC will then fill out an introductory information form. I.V. House UltraDressing (I.V. House, Inc., St. Louis, MO, USA) will be applied according to the manufacturer's instructions and secured with an anti-slip tape without the need for further taping. Catheter-induced complications such as dislodgement, phlebitis, infiltration, extravasation, catheter occlusion and folding of PVCs will be observed and recorded on the Peripheral Venous Catheter Observation Form and the effect of I.V. House UltraDressing will be evaluated.
  Interventions: Device: I.V. House UltraDressing
- Control (No Intervention): The nurse who will perform the PVC application will clean the area where the PVC will be applied with alcohol and cotton wool and leave it to dry, and the patients in both groups will be applied with a Teflon Introcan Safety I.V. Catheter (B. Braun Medical Inc. Bethlehem, PA, USA) numbered 22-24 and the clinic's routine intravenous line fixation method of fixation with a plaster will be applied. After the PVC is inserted, the introductory information form will be filled out and the duration of the stay of the PVC in the vascular access, dislodgement status and catheter-related complications such as dislodgement, phlebitis, infiltration, extravasation, catheter occlusion and folding of the PVCs will be observed and recorded on the Peripheral Venous Catheter observation form prepared by the researcher. Patients will remain in the study as long as they are hospitalized in the clinic and their PVCs are inserted. The time allocated for each patient is planned to last an average of 15 minut

INTERVENTIONS:
Device: I.V. House UltraDressing — I.V. House UltraDressing (I.V. House, Inc., St. Louis, MO, USA) will be applied according to the manufacturer's instructions and secured with an anti-slip tape without the need for further taping. It is intended to prevent complications such as catheter-related displacement, phlebitis, infiltration, extravasation, catheter occlusion, and folding of PVCs.
  Arms: I.V. House UltraDressing

SUMMARY:
Objective: This study aimed to determine the effect of applying the IV House Ultradressing catheter protector on the frequency of peripheral venous catheter (PVC) replacements and complications in patients with peripheral venous catheterization in an oncology clinic.

Materials and Methods: The research was planned as a randomized controlled experimental study. The population of the study consisted of patients hospitalized in the oncology clinic. The sample of the study was calculated based on the data from the study by Büyükyılmaz et al. (2019), which found a significant difference in the average duration of catheter-related phlebitis in the intervention group (2.10 ± 1.55 days) compared to the control group (1.27 ± 0.45 days), with an effect size of d=0.72. As a result of the sample size calculation, 32 patients were predicted for each group. Considering that 10% of patients might drop out during the study, a total of 70 patients, with 35 in each group, were decided to be included. After the catheter is inserted, patients in the intervention group will have their catheter area protected with IV House Ultradressing, while no protective measures will be applied to the control group. Both groups will be evaluated in terms of catheter duration and PVC complications. It is planned to use t-tests and chi-square tests for data analysis.

DETAILED DESCRIPTION:
The aim of this study was to determine the effect of IV House Ultradressing catheter protector application on the frequency of PVC change and complications in patients hospitalized in an oncology clinic and undergoing peripheral venous catheterization.

Research Question and Hypotheses H01: There is no difference in the frequency of PVC replacement between the IV House UltraDressing intervention group and the control group.

H02: There is no difference in PVK-related complications between the IV House UltraDressing intervention group and the control group.

H11: There is a difference in the frequency of PVK replacement between the IV House UltraDressing intervention group and the control group.

H12: There is a difference in PVK-related complications between the IV House UltraDressing intervention group and the control group.

MATERIALS AND METHODS

Type of Research

This study is planned to be conducted as a pretest-posttest, parallel group randomized controlled experimental design to evaluate the efficacy of IV House UltraDressing on the frequency of PVC change and catheter complications in patients treated in an oncology clinic. It was thought that the application of IV House UltraDressing would significantly reduce the frequency of PVC change and complications.

Population and Sample of the Study The research will be conducted with patients hospitalized in Necmettin Erbakan University Faculty of Medicine Oncology Clinic between October 2024 and March 2025. The sample size of the study was determined using the G. Power-3.1.9.2 program, with a power of 1-β=0.80 and an error level of α=0.05. Based on the data in the study of Büyükyılmaz et al. (2019), the effect size was calculated as d=0.72 based on the finding that there was a significant difference between the average duration of stay due to catheter-induced phlebitis in the intervention group (2.10 ± 1.55 days) and the average in the control group (1.27 ± 0.45 days). As a result of the sample size calculation made according to this assumption, 32 patients were predicted for each group. When it was predicted that 10% of the patients would leave the sample throughout the study, it was decided to include a total of 70 patients in the study, 35 patients in each group.

Randomization

The study group will be formed according to the inclusion and exclusion criteria. Patients who agree to participate in the study will be divided into two groups as intervention (IV House UltraDressing) and control group. The assignment of patients to the groups will be performed randomly by a statistician other than the researcher using a computer program (https://www.randomizer.org). Patients will be assigned by simple randomization method to protect confidentiality and prevent bias, and allocation to groups will be by block randomization method.

Blinding Patients will be informed about the study without disclosing which group they are in and their consent will be obtained. The researcher collecting the data for the study will be informed by telephone by an independent person after the written consent of the patients has been obtained and the pre-test data has been collected. Since the researcher manages the implementation process of the study, researcher blinding will not be possible.

The study will also be blinded in terms of statistical analysis. The data will be recorded on the computer by the researcher as group A and group B without using the terms experimental and control group. Data analyses will be performed by a statistician other than the randomizer.

Data Sources and Data Collection Method

The research data will be collected with the Introductory Information Form, which inquires the descriptive characteristics of the patients prepared by the researcher, and the PVK Follow-up Form.

Introductory Information Form: This part of the data collection form prepared by the researcher includes information such as the patient's age, gender, height, weight, hospitalization diagnosis, hospitalization date, and chronic diseases.

PVC Follow-up Form: The PNC follow-up form prepared by the researcher includes information on the date of insertion and removal of the PNC, the anatomical region where the PNC was inserted, the catheter number used, the duration of stay in the vein, the reason for changing the catheter (phlebitis, infiltration, extravasation, dislocation, catheter occlusion and catheter folding), the medications and IV fluids given, the status of blood product administration and the degree of phlebitis.

Phlebitis Assessment Scale: Phlebitis will be diagnosed with the phlebitis assessment scale developed by the Intravenous Nurses Association. The degree of phlebitis will be evaluated by measuring the width of the phlebitis area with a transparent millimeter ruler used by the investigators. The scale includes grading steps from 0 to 4 by observing the symptoms that can be seen at each stage of phlebitis.

Phlebitis with this scale:

* Grade 0: no symptoms,
* Grade 1: redness and/or pain at the catheter entry site,
* Grade 2: redness, pain and/or edema at the catheter entry site,
* Grade 3: redness, pain and/or edema at the catheter entry site, red line, palpation of the vein as a cable, Grade 4: redness, pain and/or edema at the catheter entry site, red line, palpation of the vein as a cable and longer than 2.5 cm, purulent discharge.

Research Implementation

The study will be conducted between October 2024 and March 2025. The study, which is planned as intervention and control groups, will start with the patients who have PVK implanted and who have informed that they agree to participate in the study. The data in both groups will be collected by the researcher every 24 hours and by the clinic nurses every 8 hours by interview and observation method. In the study, the duration of stay in the vein of a single catheter and newly opened catheter will be evaluated. In addition, a single vascular access will be evaluated in patients with more than one vascular access. The IV access will be performed by the nurse working in the clinic.

Intervention Group: The nurse who will perform the PVC will clean the area where the PVC will be applied with alcohol and cotton wool, let it dry and apply Teflon Introcan Safety I.V. Catheter No. 22-24 (B. Braun Medical Inc. Bethlehem, PA, USA) to the patients and apply the routine intravenous line fixation method of the clinic with a plaster. The patient with the PVC will then fill out an introductory information form. I.V. House UltraDressing (I.V. House, Inc., St. Louis, MO, USA) will be applied according to the manufacturer's instructions and secured with an anti-slip tape without the need for further taping. Catheter-induced complications such as dislodgement, phlebitis, infiltration, extravasation, catheter occlusion and folding of PVCs will be observed and recorded on the Peripheral Venous Catheter Observation Form and the effect of I.V. House UltraDressing will be evaluated.

Control Group: The nurse who will perform the PVC application will clean the area where the PVC will be applied with alcohol and cotton wool and leave it to dry, and the patients in both groups will be applied with a Teflon Introcan Safety I.V. Catheter (B. Braun Medical Inc. Bethlehem, PA, USA) numbered 22-24 and the clinic's routine intravenous line fixation method of fixation with a plaster will be applied. After the PVC is inserted, the introductory information form will be filled out and the duration of the stay of the PVC in the vascular access, dislodgement status and catheter-related complications such as dislodgement, phlebitis, infiltration, extravasation, catheter occlusion and folding of the PVCs will be observed and recorded on the Peripheral Venous Catheter observation form prepared by the researcher. Patients will remain in the study as long as they are hospitalized in the clinic and their PVCs are inserted. The time allocated for each patient is planned to last an average of 15 minutes.

Application tools

I.V. House UltraDressing: Developed by pediatric nurses Lisa Vallino and Betty Rozier in 1991, the I.V. House UltraDressing is an innovative product developed to provide, stabilize and protect long-term catheter safety. The product is a clear plastic dome that protects the catheter connection point. There is also a soft foam pad under the outer dome edge to ensure patient comfort (IV. House, Inc., St. Louis, MO, USA). The use of safe fixation methods is key in preventing complications related to PVK. Therefore, in this data collection method, in the intervention group, after filling out the introductory information form, IV. House UltraDressing will be applied to the inserted PVC and the frequency of catheter change and catheter-related complications will be evaluated and recorded in the PVC follow-up form.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria
* Hospitalized in the oncology clinic
* The one with the PVK attached,
* Volunteered to participate in the research,
* Treated in the same clinic during the study period,
* No verbal, perceptual and visual communication problems,
* 22-24 G (Blue) size catheter used,
* Between the ages of 18 and 65,
* Literate,
* Patients without scar tissue, infection, hematoma, edema at the sites to be used for PVK placement were included in the study.

Exclusion Criteria:

* - With a clotting disorder,
* Patients with problems with skin integrity or limb movement such as scar tissue, infection, hematoma, edema at the PVK site,
* Blood or blood products given through a catheter,
* Patients who wanted to leave, were referred to a different clinic or discharged during the study were excluded from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Phlebitis Follow up Form | up to 1 weeks
  The scale includes grading steps from 0 to 4, with observation of symptoms that can be seen at each stage of phlebitis.
  With this scale, phlebitis is evaluated as:
  * Grade 0: no symptoms,
  * Grade 1: redness and/or pain at the catheter entry site,
  * Grade 2: redness, pain and/or edema at the catheter entry site,
  * Grade 3: redness, pain and/or edema at the catheter entry site, red line, palpation of the vein in the form of a cable, Grade 4: redness, pain and/or edema at the catheter entry site, red line, palpation of the vein in the form of a cable and longer than 2.5 cm, purulent discharge.
PIVC Length of Stay Follow up Form | up to 1 weeks
  The purpose of this form is to determine how many days PIVC remains in the patient. The form includes the items for day 0, day 1, day 2, day 3, day 4, day 5, day 6 and day 7.
Infiltration Follow up Form | up to 1 weeks
  The purpose of this form will be used to determine infiltration. The form includes "yes" and "no" items. After the catheter is assessed by observation and palpation, the present item will be marked if there is infiltration, and the absent item will be marked if there is no infiltration.
Extravasation Follow up Form | up to 1 weeks
  The purpose of this form will be used to determine extravasation. The form includes "yes" and "no" items. After the catheter is assessed by observation and palpation, the present item will be marked if there is extravasation, and the absent item will be marked if there is no extravasation.
Occlusion Follow up Form | up to 1 weeks
  This form will be used to determine the occlusion in the PIVC.The form includes "yes" and "no" items. After the catheter is assessed by observation and palpation, the present item will be marked if there is occlusion, and the absent item will be marked if there is no occlusion.
Folding Follow up Form | up to 1 weeks
  This form will be used to determine the folding in the PIVC. The form includes "yes" and "no" items. After the catheter is assessed by observation and palpation, the present item will be marked if there is folding, and the absent item will be marked if there is no folding.
Dislocation Follow up Form | up to 1 weeks
  This form will be used to determine PIVC dislocation.The form includes "yes" and "no" items. After the catheter is assessed by observation and palpation, the present item will be marked if there is dislocation, and the absent item will be marked if there is no dislocation.

CONTACTS AND LOCATIONS:
Overall Officials: BETÜL TOSUN, DOÇ. DR., Principal Investigator — Karamanoğlu Mehmetbey University

IPD SHARING:
Plan to Share IPD: Undecided